CLINICAL TRIAL: NCT05975086
Title: Right Ventricle Dysfunction in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Shaban Abdelsalam Thabet, Resident doctor, Assiut University
Other Study IDs: RVD
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess prevalence of right ventricle dysfunction in critically ill patient. To assess impact of RV dysfunction on short term (ICU stay, hospital stay, or mortality ≤30 days) and long term outcome (>30 days).

To assess the accuracy of different parameters of RV dysfunction.

DETAILED DESCRIPTION:
1. Inclusion criteria:

   - Adult patients who admitted to critical care of Internal medicine department after obtaining consent during the period between august 2023 and august 2024.
2. Exclusion criteria:

   1. Children below 18 yr.
   2. Patients who could not be scanned within 48h after ICU admission.
3. Sample Size Calculation:

   200 patients 2.4.4 Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, ):

   Beside history and clinical examination , The following data will be obtained:

   Demographic and historical data: the patient age, sex, history of hypertension, chronic obstructive pulmonary disease, IHD, cause of critical care unit admission and indication of mechanical ventilation( PEEP).

   Clinical examination data: pulse, blood pressure, respiratory rate, temperature , BMI, and thorough chest, cardiac examination data will be obtained.

   Volume state of the patient: CVP measurement, input and output fluid chart. APACHE IV score, Use of vasopressors, Use of sedatives. Investigation : Arterial blood gas analysis, pulse oxygen saturation, CBC, and renal function test and electrolytes, serum lactate and troponin.

   12 lead ECG for RV strain patterns.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who admitted to critical care of Internal medicine department after obtaining consent during the period between august 2023 and august 2024.

Exclusion Criteria:

1. Children below 18 yr.
2. Patients who could not be scanned within 48h after ICU admission.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Adult patients who admitted to critical care of Internal medicine department after obtaining consent during the period between august 2023 and august 2024.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Impact of right ventricle dysfunction in Critically ill patients on short term and long term outcome | Baseline
  To assess prevalence of right ventricle dysfunction in critically ill patient. To assess impact of RV dysfunction on short term (ICU stay, hospital stay, or mortality ≤30 days) and long term outcome (>30 days).

SECONDARY OUTCOMES:
Impact of right ventricle dysfunction in Critically ill patients on short term and long term outcome | Baseline
  To assess prevalence of right ventricle dysfunction in critically ill patient. To assess impact of RV dysfunction on short term (ICU stay, hospital stay, or mortality ≤30 days) and long term outcome (>30 days).

REFERENCES:
- [Background] Vieillard-Baron A, Millington SJ, Sanfilippo F, Chew M, Diaz-Gomez J, McLean A, Pinsky MR, Pulido J, Mayo P, Fletcher N. A decade of progress in critical care echocardiography: a narrative review. Intensive Care Med. 2019 Jun;45(6):770-788. doi: 10.1007/s00134-019-05604-2. Epub 2019 Mar 25. PMID 30911808
- [Background] Vieillard-Baron A, Naeije R, Haddad F, Bogaard HJ, Bull TM, Fletcher N, Lahm T, Magder S, Orde S, Schmidt G, Pinsky MR. Diagnostic workup, etiologies and management of acute right ventricle failure : A state-of-the-art paper. Intensive Care Med. 2018 Jun;44(6):774-790. doi: 10.1007/s00134-018-5172-2. Epub 2018 May 9. PMID 29744563
- [Background] Vieillard-Baron A, Pinsky MR. The difficulty in defining right ventricular failure at the bedside and its clinical significance. Ann Intensive Care. 2021 Aug 5;11(1):122. doi: 10.1186/s13613-021-00912-7. No abstract available. PMID 34351534
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Vos ME, Cox EGM, Schagen MR, Hiemstra B, Wong A, Koeze J, van der Horst ICC, Wiersema R; SICS Study Group. Right ventricular strain measurements in critically ill patients: an observational SICS sub-study. Ann Intensive Care. 2022 Oct 3;12(1):92. doi: 10.1186/s13613-022-01064-y. PMID 36190597
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077